CLINICAL TRIAL: NCT02388880
Title: Physiological Effects of Intrathoracic Pressure Regulation in Patients With Decreased Cerebral Perfusion Due to Brain Injury or Intracranial Pathology (4 Hour Use)
Brief Title: Effect of Intrathoracic Pressure Regulation on Decreased Cerebral Perfusion (4hour)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than anticipated enrollment
Sponsor: Advanced Circulatory Systems (Industry)
Collaborators: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACSI 450-0003; W81XWH-12-C-0181 (Other Grant/Funding Number: United States Army Institute for Surgical Research)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-03

CONDITIONS: Head Injury; Intracranial Pathology; Compromised Cerebral Perfusion
Keywords: ITPR; CPP; TBI; traumatic brain injury; cerebral perfusion pressure; intrathoracic pressure regulator
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITPR (Experimental): Use of the ITPR for 240 minutes.
  Interventions: Device: ITPR

INTERVENTIONS:
Device: ITPR — Single use noninvasive device that is connected to a vacuum source and a means to deliver a positive pressure breath. The device generates negative pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure between the periods of positive pressure ventilations.
  Other Names: Intrathoracic Pressure Regulator; CirQlator

SUMMARY:
The purpose of the study is to evaluate the physiological response to application of the Intrathoracic Pressure Regulator (ITPR) in patients with compromised cerebral circulation. The study will evaluate the physiological response to intrathoracic pressure regulation (IPR) therapy in hemodynamically stable patients with compromised cerebral circulation who are on ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* intubated and mechanically ventilated on a volume controlled mode
* head injury or other intracranial pathology and compromised cerebral perfusion
* arterial line in place or alternative with continuous pressure monitoring
* SpO2 ≥90%
* mean arterial pressure >55
* admission to ICU or about to undergo neurosurgery with planned placement of an invasive intracranial pressure monitor
* inclusion presents no significant delays to planned emergent neurosurgery
* prior written informed consent

Exclusion Criteria:

* cardiac or pulmonary injury
* confirmed pneumothorax or hemothorax
* serious neck injury resulting in neck swelling with jugular venous compression
* evidence of ongoing uncontrolled bleeding
* respiratory disease such as COPD, interstitial lung disease, or other parenchymal or pulmonary vascular disease
* marked hypertension at time of device use defined as systolic blood pressure >180 mmHg
* congestive heart failure
* women with positive serum or urine pregnancy test or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ITPR
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ITPR
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.67 (18.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Perfusion Pressure (CPP)
Description: Change from baseline CPP compared with the CPP during use of the ITPR.
Time Frame: During 240 minutes of device use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 3
mmHg | -4.88 (6.29)

2. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: Change from baseline MAP compared with the MAP during use of the ITPR.
Time Frame: baseline to end of ITPR use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 3
mmHg | -4.08 (14.5)

3. Secondary Outcome: Intracranial Pressure (ICP)
Description: Change from baseline ICP compared with the ICP during use of the ITPR.
Time Frame: baseline to end of ITPR use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 3
mmHg | 1.05 (9.63)

4. Secondary Outcome: End-tidal Carbon Dioxide (EtCO2)
Description: Change from baseline EtCO2 compared with the EtCO2 during use of the ITPR.
Time Frame: baseline to end of ITPR use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITPR
Number analyzed (Participants) | 3
mmHg | 0.42 (7.07)

ADVERSE EVENTS:
Time Frame: Duration of device use.
Arm/Group | ITPR
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITPR (N=3)
Increase in ICP >10mmHg (Vascular disorders) | 1 (1)
Decrease in MAP >20mmHg (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITPR (N=3)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less